CLINICAL TRIAL: NCT00215228
Title: Effects of Escitalopram vs. Duloxetine on Heart Rate Variability and Autonomic Cardiovascular Control
Brief Title: Effects of Duloxetine vs. Escitalopram on Heart Rate Variability in Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00007159; 6957-05-3R0 (Other: DUMC)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2007-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Drug: duloxetine vs. escitalopram

SUMMARY:
Low heart rate variability is a marker of increased risk of cardiac mortality, and is observed in depressed coronary artery disease patients. Some antidepressants may themselves, however, decrease heart rate variability. We will test the hypothesis that greater reduction in heart rate variability will be associated with duloxetine (which has noradrenergic activity) than escitalopram (a selective serotonin reuptake inhibitor). We will also test the hypothesis that changes in heart rate variability are related to the magnitude of norepinephrine transporter occupancy.

DETAILED DESCRIPTION:
Evaluation of heart rate variability (HRV) has been shown to be a valuable tool for measuring autonomic dysfunction associated with depression and with cardiac disease. Low HRV is a marker of increased risk of cardiac mortality, and is observed in depressed coronary artery disease patients and in anxious patients post-MI. Treatment with sympathomimetic antidepressants, such as MAO inhibitors and tricyclics, reduce HRV further, and have been associated with elevated heart rate, orthostatic hypotension, and with adverse cardiac events. Although there is increasing evidence that the selective serotonin reuptake inhibitor (SSRI) class of antidepressants have minimal effects on the cardiovascular system, the case is less clear with the SNRI antidepressants which block the reuptake of both serotonin and norepinephrine. It is possible that measures of the extent of norepinephrine transporter blockade or inhibition may relate to the HRV reduction seen with noradrenergic drugs. Given these considerations, we propose a study to compare the cardiovascular profile of the SSRI escitalopram (Lexapro), with the most recently available SNRI, duloxetine, in outpatients with depression. Using HRV methodology, we will test the hypothesis that greater reduction in HRV will be associated with duloxetine than escitalopram. In addition, we will measure the magnitude of serotonin and norepinephrine transporter occupancy produced by each drug. This will allow us to examine the relationship between changes in HRV to the magnitude of transporter inhibiting effects of each drug.

ELIGIBILITY:
Inclusion Criteria:

* adults 20-60 years of age
* a primary diagnosis of depression using DSM-IV criteria
* written informed consent
* a negative serum pregnancy test for women of childbearing potential

Exclusion Criteria:

* history of cardiovascular disease
* history of hypertension
* history of bipolar disorder
* history of schizophrenia or other psychotic disorder
* alcohol or other substance abuse within the last 3 months
* history of cognitive impairment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2005-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Effect of treatment on heart rate variability

SECONDARY OUTCOMES:
Effect of treatment on affective variables (depression, anxiety, stress reactivity)
Effect of treatment on neurotransmitter transporter occupancy

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, M.D., Ph. D, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States